CLINICAL TRIAL: NCT04470076
Title: Neoadjuvant Afatinib Combination With Chemotherapy for Stage Ⅱa-Ⅲb Non-small Cell Lung Cancer With Epidermal Growth Factor Receptor Activating Mutation
Brief Title: Neoadjuvant Afatinib Combination With Chemotherapy for Stage Ⅱa-Ⅲb NSCLC With EGFR Activating Mutation
Acronym: Neoafa
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.XXWK002
Record Dates: First submitted 2020-07-03; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Non Small Cell Lung Cancer; Surgery; EGFR Activating Mutation; Chemotherapy; EGFR TKI
Keywords: neoadjuvant therapy; dynamic 18F-FDG PET/CT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine; Cisplatin; Carboplatin; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant afatinib combination with chemotherapy (Experimental): Neoadjuvant treatment (chemotherapy+afatinib) will start within 1-3 days from enrollment/randomisation. 3 cycles will be administered at 21-day (+/- 3 days) intervals (QW3) prior to surgery. Before surgery a tumor assessment (including dynamic 18F-FDG PET/CT) will be done. Patients must leave the study if there is evidence of progression. Patients with stable disease or partial response may be considered for surgery.
  Surgery: Surgery must be done within the 3rd-4th week (+7 days) from day 21 cycle 3 of neoadjuvant treatment (day 42-49 after day 1 of cycle 3) Adjuvant treatment (afatinib): Patients that are R0 confirmed by surgical pathology evaluation will receive the first adjuvant administration within the first week (+ 7 days) from surgery and up to 2 years.
  Interventions: Drug: Neoadjuvant treatment: Afatinib, pemetrexed, gemcitabine, cisplatin, carboplatin; Procedure: Surgical treatment; Drug: Adjuvant treatment:afatinib

INTERVENTIONS:
Drug: Neoadjuvant treatment: Afatinib, pemetrexed, gemcitabine, cisplatin, carboplatin — ① Eligible patients with non-squamous cell lung cancer will receive pemetrexed 500mg/m2, IV on day 1 and cisplatin 75mg/m2 or carboplatin area under curve (AUC) =5, on day 1 of a 3-week schedule for 3 cycles.
  ② Eligible patients with squamous cell lung cancer will receive gemcitabine 1250mg/m2 IV on day 1 and day 8, and cisplatin 75mg/m2 or carboplatin AUC =5 on day 1 of a 3-week schedule for 3 cycles .
  ③Patient will take afatinib at dosage of 30mg per day 48 hours after chemotherapy and will stop 24 hours before next cycle of chemotherapy.
Procedure: Surgical treatment — The patients who respond to neoadjuvant treatment (CR+PR) and the patients who do not respond to therapy but could still undergo surgery (SD and PD) will receive radical lung resection 3-4 weeks later after neoadjuvant.
Drug: Adjuvant treatment:afatinib — The CR, PR and SD patients who have been treated surgically will take afatinib at a dosage of 30mg per day for 2 year.

SUMMARY:
The recommended adjuvant therapy for stage Ⅱa-Ⅲb Non-small cell lung cancer (NSCLC) were perioperative chemotherapy. The adjuvant or neoadjuvant chemotherapy for early stage lung cancer improved about 5% 5-year survival. As for advanced NSCLC with epidermal growth factor receptor (EGFR) activating mutation, epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) combination with chemotherapy had improved progression-free survival (PFS) compared with EGFR-TKI alone. We propose this trial of Neoadjuvant Afatinib Combination With Chemotherapy for Stage Ⅱa-Ⅲb NSCLC With EGFR Activating Mutation, which would maximize benefit early in a patient's treatment course. At the same time, dynamic 18F-2-fluoro-2-deoxy-D-glucose positron emission tomography (18F-FDG PET) was used to evaluate the standardized uptake value (SUV) and uptake rate constant (Ki) changes of lesions before and after treatment, so as to accurately and quantitatively monitor the tumor response of different therapy.

DETAILED DESCRIPTION:
The prognosis of stage Ⅱa-Ⅲb Non-small cell lung cancer (NSCLC) was worse, with 5-year survival rate between 26%-60%. The recommended adjuvant therapy for stage Ⅱa-Ⅲb NSCLC were adjuvant or neoadjuvant chemotherapy. As for advanced NSCLC with EGFR activating mutation, EGFR-TKI combination with chemotherapy had improved survival compared with EGFR-TKI alone. The Chinese Thoracic Oncology Group-1103 (CTONG-1103) trial showed that neoadjuvant erlotinib has better PFS than neoadjuvant chemotherapy.

The investigators propose that neoadjuvant EGFR-TKI combination with chemotherapy for stage Ⅱa-Ⅲb NSCLC with EGFR activating mutation might have better pathological response and disease-free survival (DFS) than chemotherapy alone, and maximize benefit early in a patient's treatment course. At the same time, dynamic 18F-2-fluoro-2-deoxy-D-glucose positron emission tomography (18F-FDG PET) was used to evaluate the standardized uptake value (SUV) and uptake rate constant (Ki) changes of lesions before and after treatment, so as to accurately and quantitatively monitor the tumor response of different therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC, performed on a biopsy that occurred within the last 60 days
* Computed tomography (CT) or PET-CT within the last 30 days showing radiographic stage Ⅱa to Ⅲb lung cancer (mediastinal staging biopsy is allowed but not required) by the American Joint Committee on Cancer (AJCC) 8th edition
* Deemed surgically resectable by a senior thoracic surgeon
* Age≥18 years, and ≤75 years
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the investigator
* Adequate tissue specimens for correlative biomarker analysis. The patient should be willing to provide tissue from a newly obtained biopsy of a tumor lesion and surgical resected tumor lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy or surgical procedures to NCI CTCAE version (v)5.0 grade 1
* Be willing and able to provide written informed consent for the trial
* Absolute neutrophil count (ANC) >= 1500 cells/ microlitre(uL) (within 10 days prior to the start of trial treatment)
* Platelets >= 100 000 cells/uL (within 10 days prior to the start of trial treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks) (within 10 days prior to the start of trial treatment)
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance, glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl) >= 30 mL/min for patients with creatinine levels > 1.5 x institutional ULN (within 10 days prior to the start of trial treatment)
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN (within 10 days prior to the start of trial treatment)
* Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 x ULN (=< 5 x ULN for patients with liver metastases) (within 10 days prior to the start of trial treatment)
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of trial treatment)
* Activated partial thromboplastin time (aPTT)/PTT =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of trial treatment)
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Male and female patients of childbearing potential must be willing to use an adequate method of contraception as outlined, for the course of the trial through 120 days after the last dose of trial drug

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient

Exclusion Criteria:

* Any approved anticancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 years prior to initiation of study treatment; however, the following are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy > 1 week prior to Cycle 1, Day 1 (herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to Cycle 1, Day 1)
* Malignancies other than the disease under study within 3 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0, prostate cancer with Gleason score ≤ 6, and prostate-specific antigen (PSA) ≤ 10 mg/mL, etc.)
* Patients who are receiving any other investigational agents concurrently.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to afatinib, cisplatin, carboplatin, pemetrexed or gemcitabine.
* Patients with active hepatitis B or C infections or a history of HIV infection.

  * Patients with past or resolved hepatitis B infection, defined as having a negative hepatitis B surface antigen (HBsAg) test and a positive for the antibody test to detect antibodies to hepatitis B core antigen (anti-HBc) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection including tuberculosis (TB), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible.
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1 Received oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live, attenuated vaccine will be required during the study
* Pregnant women
* History of interstitial lung disease or pneumonitis of any cause
* Is ineligible for an operation based on medical or oncologic contraindications to surgery
* Is currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of trial treatment

  * Note: Patients who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-10 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Major pathological response | up to 12 weeks; analysis of surgical resected tumor samples after neoadjuvant therapy
  10% or less residual viable tumor cells
Objective response rate | up to 12 weeks; after neoadjuvant therapy
  Image assessment of tumor response according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression free survival | Pts after surgery will receive long-term follow-up including chest CT scan, abdominal ultrasound every 3 months, brain MRI every 6 months, bone scan (ECT) every 12 months for up to 3 years
  Time from enrollment to disease progression or death from any cause, whichever occurred first
Overall survival | up to 100 months
  From date of randomization until the date of date of death from any cause, whichever came first, assessed up to 100 months
R0 resection | up to 12 weeks; analysis of surgical resected tumor samples
  the proportion of patients with negative surgical margin and no residual found under microscope after resection in all patients who have completed the treatment
Treatment related adverse events | 12 weeks
  the number of adverse events related to afatinib or platinum-based chemotherapy as evaluated according to CTCAE v4.0.
standardized uptake value (SUV) changes | up to 12 weeks; before and after neoadjuvant therapy
  standardized uptake value (SUV) changes before and after neoadjuvant therapy
uptake rate constant (Ki) changes | up to 12 weeks; before and after neoadjuvant therapy
  uptake rate constant (Ki) changes before and after neoadjuvant therapy

IPD SHARING:
Plan to Share IPD: Undecided
The researchers will consider whether individual participant data (IPD) is available to other researchers only after the paper is published